CLINICAL TRIAL: NCT06360705
Title: An Exploratory Open Label Trial of StrataMGT for the Treatment of Vulvar Lichen Sclerosus
Brief Title: StrataMGT for the Treatment of Vulvar Lichen Sclerosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Vulvovaginal Disorders (Other)
Collaborators: Stratpharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVVD003
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Vulvar Lichen Sclerosus
MeSH Terms: conditions — Vulvar Lichen Sclerosus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Exploratory Open Label (Experimental): Experimental: StrataMGT
  Interventions: Device: StrataMGT

INTERVENTIONS:
Device: StrataMGT — StrataMGT® is a semi-permeable, non-resorbable and self-drying gel. StrataMGT® contains no steroids, hormones, alcohol, parabens or fragrances. StrataMGT® gel is bacteriostatic, inert, and is manufactured in compliance with good manufacturing practices (GMPs), 21CFR210 and 211.

SUMMARY:
This study is designed to evaluate the efficacy and safety of StrataMGT for the treatment of vulvar lichen sclerosus.

DETAILED DESCRIPTION:
This will be an exploratory open label study to evaluate the efficacy and safety of StrataMGT for the treatment of vulvar lichen sclerosus. 5 patients with a diagnosis of biopsy proven vulvar lichen sclerosus will be recruited from one center. This study will consist of a two-week screening period and an 8-week treatment period. At the beginning of the screening period, a vulvoscopy will be performed at the screening visit and after the 8-week treatment period to rule out vulvar intraepithelial neoplasia (VIN) or carcinoma. All patients will have a 4mm punch biopsy at screening (week 0) and after 8 weeks of treatment (week 10).

The primary efficacy variable will be performed by a dermatopathologist who will evaluate the inflammatory infiltration on biopsy specimens obtained during the screening period and after treatment at the Week 10 visit (0 to 3 scale).

Secondary efficacy endpoints will be change in score on the Vulvar Quality of Life Index (VQLI), the Skindex 29, and the Clinical Lichen Sclerosus Scoring Scale (CLISSCO).

ELIGIBILITY:
Inclusion criteria:

Subjects to be included are those:

* Female, 18 years or older.
* With a diagnosis of biopsy proven vulvar lichen sclerosus.
* Signed written informed consent.
* Willingness and ability to comply with the study requirements.
* Subject must have a score of 16 or greater in the VQLI at screening.
* Women must have a culture negative for candidiasis or bacterial vaginosis at screening. Subjects who screen positive for either candidiasis or bacterial vaginosis at the screening visit may be treated and retested and may participate if the confirmatory test after treatment is negative. Any vulvovaginal infections during participation in the study will be considered an adverse event. The subject will then stop the study IP and will be treated for the infection and may resume use of the IP 3 days after the last dose of medication for the infection. Participants will be discontinued from the study if participants have two infections during the study.

Exclusion criteria:

Subjects to be excluded are those:

* Who have received systemic immunosuppressants (e.g. corticosteroids) within 12 weeks prior to participation in the study.
* Who have been treated with topical therapy (e.g., topical corticosteroids, topical calcineurin inhibitors, topical estrogen, topical testosterone) at the affected area within 12 weeks prior to participation in the study.
* Who use topical emollients, lubricants (other than for penetrative intercourse),or any other topical products for symptom control at the affected area within 4 weeks prior to participation in the study.
* Prior history of, or active Vulvar Intraepithelial Neoplasia (VIN) or vulvar carcinoma.
* Who are immunocompromised (e.g., lymphoma, AIDS, Wiskott-Aldrich Syndrome) or have an uncontrolled malignant disease.
* Who suffer from systemic or generalized infections (bacterial, viral or fungal).
* Who have been diagnosed with lichen planus, psoriasis, candidiasis, intraepithelial neoplasia, or carcinoma of the vulva.
* Who had received an investigational drug within four weeks prior to the study or who intend to use other investigational drugs during the course of this study.
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study.
* Who have a history of substance abuse or any factor, which limits the subject's ability to cooperate with the study procedures.
* Who are uncooperative, known to miss appointments (according to subjects' records) and are unlikely to follow medical instructions or are not willing to attend regularly scheduled visits.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cis-gendered female patients
Enrollment: 5 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Histopathologic Inflammation | 10 weeks
  Histopathologic inflammation that occurs with lichen sclerosus will be assessed by a dermatopathologist on 4mm punch biopsies performed during the screening visit (Week 0) and at the Week 10 visit using the following clinical scoring scale. The scale is from 0-3, 0 being no disease of inflammation and 3 being severe disease or inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Centers for Vulvovaginal Disorders, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No